CLINICAL TRIAL: NCT01554033
Title: Study of Huntington Patients in Connection With European Huntington's Disease Network (EHDN).
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: European Huntington's Disease Network (Network)
Responsible Party: Sponsor
Other Study IDs: H-0902-023-271
Record Dates: First submitted 2012-03-11; First posted 2012-03-14 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Huntington Disease
Keywords: European Huntington's Disease Network; Huntington patients in KOREA
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum-60ml urine-60ml Formation study of Lymphoblast and diagnosis of a Huntington gene
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Huntington's disease patients: Huntington's disease patients and his(/her) family
- age-sex matched control: age-sex matched control about huntington patients

SUMMARY:
REGISTRY is a multi-centre, multi-national, prospective, observational study of Huntington's disease (HD) with a control group of volunteers. It is an open-ended study which will include as many eligible participants as willing to participate. The goal of the project is to collect longitudinal data on the phenotypical characteristics of HD gene mutation carriers regardless of whether they display clinical symptoms and signs of the disease and of individuals who are part of an HD family (irrespective of their mutation carrier status), in order to:

* obtain natural history data on a wide spectrum of HD mutation carriers and individuals who are part of an HD family
* relate phenotypical characteristics

  * with genetic factors ('genetic modifiers')
  * with data derived from the study of body fluids (blood, urine - 'wet biomarker') and
  * imaging data ('dry biomarker')
* expedite identification and recruitment of participants for clinical trials
* develop and validate sensitive and reliable outcome measures for detecting onset and change over the natural course of premanifest and manifest HD which may also be potential outcome measures for use in future clinical trials and clinical care.
* plan for future research studies (observational and interventional trials aimed at better symptom control or aimed at slowing or postponing the onset and progression of HD).

DETAILED DESCRIPTION:
To collect prospective data on the phenotypical characteristics of HD mutation carriers regardless of whether they display clinical symptoms and signs of HD and of individuals who are part of an HD family (irrespective of their mutation carrier status), in order to;

* obtain natural history data on a wide spectrum of HD patients, HD mutation carriers and individuals who are part of an HD family
* relate phenotypical characteristics with

  * genetic factors ('genetic modifiers'),
  * data derived from the study of body fluids (blood, urine - 'wet biomarker') and
  * imaging data ('dry biomarker')
* expedite identification and recruitment of participants for clinical trials
* develop and validate sensitive and reliable outcome measures for detecting onset and change over the natural course of premanifest and manifest HD, and which may also be potential outcome measures for use in future clinical trials and clinical care.
* plan for future research studies (observational and interventional trials aimed at better symptom control or aimed at slowing or postponing the onset and progression of HD).

To achieve these objectives, participants are asked to donate biosamples (blood and urine) for studies to identify genetic modifiers of HD and to establish and validate biological markers tracking the progressive course of HD; in this context a family history is requested as well in order to understand the relationships of clinical data sets and biosamples from related donors. In addition, non-mutation carrying family members of participants are asked to consider donating biosamples to serve as controls.

ELIGIBILITY:
Inclusion Criteria:

The following individuals may be eligible to participate

* Individuals, confirmed HD mutation carrier
* Manifest HD, without CAG testing
* HD family member at-risk, without CAG testing
* HD family member, non-HD mutation carrier
* REGISTRY-CONTROL participants: companion/individual without HD history
* REGISTRY-COMPANION (any of the above). Participants may be male or female and of any age. All participants must be able to provide consent for themselves, have a parent/guardian who can provide parental permission, or have an authorised legal representative who can provide consent.

Exclusion Criteria:

* Participants who are unable to understand the study protocol or unable to give informed consent, and have no legal representative.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Manho, MD, PhD, Study Chair — Department of Neurology, Seoul National University Hospital
Locations (1):
- Department of Neurology, Seoul National University Hospital, Seoul, Seoul, South Korea